CLINICAL TRIAL: NCT02230579
Title: A Single Centre, Two-part, Double-blind, Randomized, Placebo-controlled Phase I Study to Investigate the Safety, Tolerability, and Pharmacokinetic Profile of Ascending Doses of MMV390048 in Healthy Adult Volunteers
Brief Title: Phase I Study of Ascending Doses of MMV390048 in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: University of Cape Town (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MMV_MMV390048_14_01
Record Dates: First submitted 2014-08-29; First posted 2014-09-03 (Estimated); Results first posted 2018-10-29 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2018-02

CONDITIONS: Malaria
Keywords: safety; tolerability; malaria
MeSH Terms: conditions — Malaria | interventions — MMV390048

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Cohort SAD1 Fasted (Experimental): Five fasted cohorts will receive a single, ascending dose of MMV390048. The starting dose will be 5mg. Cohort SAD6 will receive a single dose in a fed state
  Interventions: Drug: MMV390048 5mg; Drug: Placebo to match MMV390048
- Cohort SAD2 Fasted (Experimental): Five fasted cohorts will receive a single, ascending dose of MMV390048. The starting dose will be 5mg. Cohort SAD6 will receive a single dose in a fed state
  Interventions: Drug: MMV390048 20mg; Drug: Placebo to match MMV390048
- Cohort SAD3 Fasted (Experimental): Five fasted cohorts will receive a single, ascending dose of MMV390048. The starting dose will be 5mg. Cohort SAD6 will receive a single dose in a fed state
  Interventions: Drug: MMV390048 40mg; Drug: Placebo to match MMV390048
- Cohort SAD4 Fasted (Experimental): Five fasted cohorts will receive a single, ascending dose of MMV390048. The starting dose will be 5mg. Cohort SAD6 will receive a single dose in a fed state
  Interventions: Drug: MMV390048 80mg; Drug: Placebo to match MMV390048
- Cohort SAD5 Fasted (Experimental): Five fasted cohorts will receive a single, ascending dose of MMV390048. The starting dose will be 5mg. Cohort SAD6 will receive a single dose in a fed state
  Interventions: Drug: MMV390048 120mg; Drug: Placebo to match MMV390048
- Cohort SAD6 Fed (Experimental): Cohort SAD6, reusing volunteers from one of the previous cohorts, will receive a single dose in a fed state to evaluate the effect of food on the pharmacokinetics and tolerability
  Interventions: Drug: MMV390048 40mg; Drug: Placebo to match MMV390048

INTERVENTIONS:
Drug: MMV390048 5mg — Supplied as "powder in bottle" formulation for reconstitution pre-dose
  Other Names: MMV390048
  Arms: Cohort SAD1 Fasted
Drug: MMV390048 20mg — Supplied as "powder in bottle" formulation for reconstitution pre-dose.
  Other Names: MMV390048
  Arms: Cohort SAD2 Fasted
Drug: MMV390048 40mg — Supplied as "powder in bottle" formulation for reconstitution pre-dose
  Other Names: MMV390048
  Arms: Cohort SAD3 Fasted; Cohort SAD6 Fed
Drug: MMV390048 80mg — Supplied as "powder in bottle" formulation for reconstitution pre-dose
  Other Names: MMV390048
  Arms: Cohort SAD4 Fasted
Drug: MMV390048 120mg — Supplied as "powder in bottle" formulation for reconstitution pre-dose
  Other Names: MMV390048
  Arms: Cohort SAD5 Fasted
Drug: Placebo to match MMV390048 — Supplied as "powder in bottle" formulation for reconstitution pre-dose
  Other Names: Placebo

SUMMARY:
This is a first-in-human study of MMV390048. The study will evaluate the safety, tolerability and pharmacokinetic properties of escalating single and multiple doses of MMV390048 when administered to healthy male volunteers and female volunteers of non-childbearing potential.

In addition, the effect of food on the pharmacokinetics and tolerability of MMV390048 will be investigated.

DETAILED DESCRIPTION:
The study is a single centre, double-blind, randomised, placebo-controlled, ascending dose study in healthy male and female volunteers (of non-childbearing potential) aged 18 to 55 years.

The study will be divided into two parts. The first part will comprise up to seven fasted cohorts (8 to 10 volunteers in each) that will receive a single, ascending dose (SAD) of MMV390048 to assess its safety, tolerability and pharmacokinetic profile. The starting dose administered to the first cohort will be 5 mg. An additional cohort (cohort 8, re-using volunteers from one of the previous cohorts) will receive a single dose of MMV390048 in a fed state to evaluate the effect of food on the pharmacokinetics and tolerability of the compound.

The data obtained from each cohort during the SAD part of the study will undergo a formal review by the Safety Review Team (SRT). Should the safety profile of the compound be deemed acceptable, and the pharmacokinetic parameters indicate that acceptable levels of the drug to elicit a pharmacodynamic response can be achieved in human plasma, the study will then proceed to the second part.

During the second part of the study volunteers will receive multiple, ascending doses (MAD) of MMV390048 to assess the pharmacokinetics, safety and tolerability following multiple oral doses. Up to three cohorts of eight volunteers each will be enrolled into this part of the study. Each volunteer will receive three consecutive daily doses of MMV390048.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* Male and female (of non-childbearing potential); age 18 to 55 years, in good health as determined by past medical history, physical examination, vital signs, electrocardiogram, and laboratory tests at screening
* Hematology, clinical chemistry and urinalysis results at screening that are within the local laboratory reference range or, if outside the range, not clinically significant. AST, ALT, lactate dehydrogenase, total bilirubin, haptoglobin and hemoglobin must be within the normal reference ranges
* Body weight at least 50kg and body mass index within 18 to 32kg/m2
* Good peripheral venous access
* Able to communicate well with the investigator, to understand and comply with the requirements of the study
* Agree to stay in contact with the study site for the duration of the study, provide updated contact information as necessary, and have no current plans to move away from the study area for the duration of the study

Exclusion Criteria:

* Any acute illness upon admission to the unit on Day -1 or prior to dosing on Day 1
* Use of any other investigational drug within 30 days or five half-lives (whichever is longer) prior to the first dose of MMV390048
* history of hypersensitivity to any drugs
* history of anaphylaxis or severe allergic reaction
* Resting vital signs at either screening or baseline outside the defined ranges
* Orthostatic changes in blood pressure and heart rate measurements greater than: 20 mmHg drop in systolic blood pressure; 10 mmHg drop in diastolic blood pressure; 20 beats per minute increase in heart rate
* history of clinically significant ECG abnormalities, or any of the defined ECG abnormalities at either screening or baseline
* History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past five years, regardless of whether there is evidence of local recurrence or metastases
* Pregnant or nursing (lactating) women
* Women of child-bearing potential
* males physiologically capable of conceiving offspring UNLESS the volunteer agrees to use condoms and ensure that his partner(s) is either not of child-bearing potential or uses a highly effective method of contraception for the entire duration of the study and for twelve weeks following the last study drug administration
* Smokers (use of tobacco products in the previous three months)
* Use of any prescription drugs, herbal supplements, over--the--counter medication or dietary supplements (vitamins included) within four weeks prior to initial dosing
* Intake of grapefruit, grapefruit juice or other products containing grapefruit within 28 days of the first drug administration of the study drug
* Excessive intake of caffeine drinks or energy drinks within 48 hours before admission defined as more than three 250 ml cups of coffee a day
* Donation or loss of 400 ml or more of blood within eight weeks prior to screening or initial dosing
* Plasma donation (>100 ml) within 60 days prior to first dosing
* Hemoglobin levels below 12.5 g/dl (males) or 11.5 g/dl (females) at screening
* Haptoglobin levels outside the reference range
* Positive direct anti-globulin test
* Liver enzymes other than ALT, AST and lactate dehydrogenase elevated ≥1.5 x ULN within two weeks prior to initial dosing
* history of autonomic dysfunction within 3 years and/or recurrent history
* History of immunodeficiency diseases, including a confirmed positive HIV test result
* Positive Hepatitis B surface antigen or Hepatitis C antibody test result
* History of recurrent infection
* history of endocrine disease, in particular adrenal disorders such as Cushing's syndrome or Addison's disease, or diabetes mellitus
* history of Gilbert's Syndrome
* history of photosensitivity
* history of any food allergy
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of drugs, or which may jeopardise the safety of the volunteer or the objectives of the study
* History or presence of impaired renal function as indicated by clinically significantly abnormal creatinine or urea values, or abnormal urinary constituents
* History of drug or alcohol abuse within the 12 months prior to dosing, or evidence of such abuse as indicated by the tests and laboratory assays at screening and/or baseline
* Any clinically significant mental disorder that could limit the validity of informed consent or the volunteer's ability to comply with protocol requirements

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2014-05; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Barnes, Prof, Principal Investigator — University of Cape Town
Locations (1):
- Cinical Pharmacology, University of Cape Town, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sinxadi P, Donini C, Johnstone H, Langdon G, Wiesner L, Allen E, Duparc S, Chalon S, McCarthy JS, Lorch U, Chibale K, Mohrle J, Barnes KI. Safety, Tolerability, Pharmacokinetics, and Antimalarial Activity of the Novel Plasmodium Phosphatidylinositol 4-Kinase Inhibitor MMV390048 in Healthy Volunteers. Antimicrob Agents Chemother. 2020 Mar 24;64(4):e01896-19. doi: 10.1128/AAC.01896-19. Print 2020 Mar 24. PMID 31932368

RESULTS

PARTICIPANT FLOW:
Recruitment Details: For the purposes of this study, subjects that were re-used in SAD6 were treated as separate subjects, i.e. the entire trial population comprised 48 subjects, eight subjects in 6 cohorts.
Groups:
- Cohort SAD1 Fasted: 5mg of MMV390048: Single administration, supplied as "powder in bottle" formulation for reconstitution pre-dose
  Placebo: Single administration, supplied as "powder in bottle" formulation for reconstitution pre-dose
- Cohort SAD2 Fasted: 20mg of MMV390048: Single administration, supplied as "powder in bottle" formulation for reconstitution pre-dose
  Placebo: Single administration, supplied as "powder in bottle" formulation for reconstitution pre-dose
- Cohort SAD3 Fasted: 40mg of MMV390048: Single administration, supplied as "powder in bottle" formulation for reconstitution pre-dose
  Placebo: Single administration, supplied as "powder in bottle" formulation for reconstitution pre-dose
- Cohort SAD4 Fasted: 80mg of MMV390048: Single administration, supplied as "powder in bottle" formulation for reconstitution pre-dose
  Placebo: Single administration, supplied as "powder in bottle" formulation for reconstitution pre-dose
- Cohort SAD5 Fasted: 120mg of MMV390048: Single administration, supplied as "powder in bottle" formulation for reconstitution pre-dose
  Placebo: Single administration, supplied as "powder in bottle" formulation for reconstitution pre-dose
- Cohort SAD6 Fed: Reusing volunteers from one of the previous cohorts, will receive a single dose in a fed state to evaluate the effect of food on the pharmacokinetics and tolerability.
  40mg of MMV390048: Single administration, supplied as "powder in bottle" formulation for reconstitution pre-dose
  Placebo: Single administration, supplied as "powder in bottle" formulation for reconstitution pre-dose
- Placebo: Placebo to match MMV390048: Single administration, supplied as "powder in bottle" formulation for reconstitution pre-dose Two volunteers within each cohort (SAD1 to SAD6) were scheduled to receive placebo in a double blind manner.
Period: Overall Study
Arm/Group | Cohort SAD1 Fasted | Cohort SAD2 Fasted | Cohort SAD3 Fasted | Cohort SAD4 Fasted | Cohort SAD5 Fasted | Cohort SAD6 Fed | Placebo
Started | 6 | 6 | 6 | 6 | 6 | 6 | 12
Completed | 6 | 6 | 6 | 6 | 6 | 6 | 12
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort SAD1 Fasted: 5mg of MMV390048: Single administration, supplied as "powder in bottle" formulation for reconstitution pre-dose
- Cohort SAD2 Fasted: 20mg of MMV390048: Single administration, supplied as "powder in bottle" formulation for reconstitution pre-dose
- Cohort SAD3 Fasted: 40mg of MMV390048: Single administration, supplied as "powder in bottle" formulation for reconstitution pre-dose
- Cohort SAD4 Fasted: 80mg of MMV390048: Single administration, supplied as "powder in bottle" formulation for reconstitution pre-dose
- Cohort SAD5 Fasted: 120mg of MMV390048: Single administration, supplied as "powder in bottle" formulation for reconstitution pre-dose
- Cohort SAD6 Fed: Cohort SAD6, reusing volunteers from previous cohorts, will receive a single dose in a fed state to evaluate the effect of food on the pharmacokinetics and tolerability
  40mg of MMV390048: Single administration, supplied as "powder in bottle" formulation for reconstitution pre-dose
- Total: Total of all reporting groups
Arm/Group | Cohort SAD1 Fasted | Cohort SAD2 Fasted | Cohort SAD3 Fasted | Cohort SAD4 Fasted | Cohort SAD5 Fasted | Cohort SAD6 Fed | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 48
Age, Continuous [Mean (Full Range); unit: years] | 29.3 [19 to 44] | 34 [24 to 51] | 37 [29 to 49] | 30 [21 to 51] | 23.7 [19 to 30] | 34 [20 to 50] | 32.7 [19 to 50] | 31.7 [19 to 51]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2 | 1 | 0 | 2 | 1 | 8
  Male | 6 | 4 | 4 | 5 | 6 | 4 | 11 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 4 | 4 | 4 | 6 | 4 | 9 | 35
  White | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 2 | 2 | 0 | 2 | 2 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Subject will be in-house up to D3, and then have a follow up visit at the site on D5, 7, 10, 14, 19, 26, 29 or longer according to half life
Time Frame: up to D29 or longer according to half life
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort SAD1 Fasted | Cohort SAD2 Fasted | Cohort SAD3 Fasted | Cohort SAD4 Fasted | Cohort SAD5 Fasted | Cohort SAD6 Fed | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 12
Participants | 4 | 5 | 5 | 6 | 6 | 6 | 11

2. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) of MMV390048
Description: Pk blood collection - additional PK point may be planned final visit depending on emerging PK data, unnecessary PK points could be eliminated for the latter cohorts Investigate the effect of food on the pharmacokinetic and tolerability of the investigational drug in cohort 4 and 8
Time Frame: 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 96, 144, 216, 312, 432, 600, 672 hours post-dose
Population: One subject (SAD5 120 mg) was excluded from the PK analysis population due to concomitant use of prohibited medications known to produce drug-drug interactions with pharmacokinetic consequences.
Measure: Median (Full Range); unit: h*ng/mL
Arm/Group | Cohort SAD1 Fasted | Cohort SAD2 Fasted | Cohort SAD3 Fasted | Cohort SAD4 Fasted | Cohort SAD5 Fasted | Cohort SAD6 Fed
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 6
h*ng/mL | 2136.9 [903.1 to 3718.7] | 32727.2 [24895.2 to 38914.3] | 21050.7 [6325.4 to 37934.6] | 58668.2 [40246 to 125655.1] | 156036.2 [13053 to 208989.4] | 29004.6 [15775.1 to 72735.3]

3. Secondary Outcome: Determine ex Vivo Efficacy (IC50)
Description: Blood collection to determine efficacy of investigational drug against parasites using an ex vivo malaria assay - this was done only for cohort 3 The experimentally obtained bioassay IC50 values were determined and compared to IC50 obtained with reference serum sample spiked with a known amount of MMV390048 titrated into the P. falciparum assay.
Time Frame: up to 144 hr post dose
Population: Samples received from the remaining participants were not processed due to the fact that they were either placebo samples, or failed to reach the pre-determined in vitro IC50 of MMV390048.
Measure: Mean (Full Range); unit: ng/ml
Arm/Group | Cohort SAD1 Fasted | Cohort SAD2 Fasted | Cohort SAD3 Fasted | Cohort SAD4 Fasted | Cohort SAD5 Fasted | Cohort SAD6 Fed
Number analyzed (Participants) | 0 | 0 | 2 | 0 | 0 | 0
ng/ml |  |  | 9.475 [9.1 to 9.85] |  |  |

4. Primary Outcome: Half-life of MMV390048
Description: Pk blood collection Investigate the effect of food on the pharmacokinetic and tolerability of the investigational drug in cohort 4 and 8
Time Frame: 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 96, 144, 216, 312, 432, 600, 672 hours post-dose
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort SAD1 Fasted | Cohort SAD2 Fasted | Cohort SAD3 Fasted | Cohort SAD4 Fasted | Cohort SAD5 Fasted | Cohort SAD6 Fed
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 6
hours | 163.1 [86.9 to 297.0] | 326.1 [221.6 to 348.0] | 192.6 [84.2 to 486.2] | 200.3 [154.1 to 457.1] | 252.3 [132.5 to 263.5] | 210.8 [111.3 to 461.1]

ADVERSE EVENTS:
Arm/Group | Cohort SAD1 Fasted | Cohort SAD2 Fasted | Cohort SAD3 Fasted | Cohort SAD4 Fasted | Cohort SAD5 Fasted | Cohort SAD6 Fed | Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 1/6 | 0/6 | 0/12
Other Adverse Events (participants affected / at risk) | 4/6 | 5/6 | 5/6 | 6/6 | 6/6 | 6/6 | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort SAD1 Fasted (N=6) | Cohort SAD2 Fasted (N=6) | Cohort SAD3 Fasted (N=6) | Cohort SAD4 Fasted (N=6) | Cohort SAD5 Fasted (N=6) | Cohort SAD6 Fed (N=6) | Placebo (N=12)
generalised myoclonus (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort SAD1 Fasted (N=6) | Cohort SAD2 Fasted (N=6) | Cohort SAD3 Fasted (N=6) | Cohort SAD4 Fasted (N=6) | Cohort SAD5 Fasted (N=6) | Cohort SAD6 Fed (N=6) | Placebo (N=12)
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Diziness (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 2 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Palpitation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Medical device site reaction (Infections and infestations) | 3 | 0 | 1 | 5 | 3 | 5 | 5
Influenza like illness (General disorders) | 0 | 2 | 2 | 2 | 0 | 1 | 2
Headache (General disorders) | 0 | 1 | 2 | 1 | 1 | 1 | 1
Blood CK increased (Blood and lymphatic system disorders) | 0 | 0 | 3 | 1 | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1
Contusion (General disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Furuncle (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Thermal burn (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No